CLINICAL TRIAL: NCT02803788
Title: Comparative Study of Antiemetic Effect of Ramosetron With Combination of Ondansetron and Dexamethasone in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Post-operative Nausea Vomiting in Laparoscopic Cholecystectomy
Acronym: PONV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Government Medical College, Haldwani (Other)
Responsible Party: Principal Investigator, Dr Shagufta Ansari, COMPARATIVE STUDY OF ANTIEMETIC EFFECT OF RAMOSETRON WITH COMBINATION OF ONDANSETRON AND DEXAMETHASONE IN PATIENT UNDERGOING LAPAROSCOPIC CHOLECYSTECTOMY, Government Medical College, Haldwani
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202/GMC/IEC/04/2014
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: ramosetron, ondansetron, dexamethasone,
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — ramosetron; Ondansetron; Dexamethasone; Antiemetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group O (Active Comparator): this group will receive inj. ondansetron 4mg iv stat and inj. dexamethasone 8mg iv stat just before extubation.
  Interventions: Drug: ramosetron, ondansetron, dexamethasone
- Group R (Experimental): this group will receive inj. ramosetron 0.3mg iv stat just before extubation.
  Interventions: Drug: ramosetron, ondansetron, dexamethasone

INTERVENTIONS:
Drug: ramosetron, ondansetron, dexamethasone — prevention of post-operative nausea vomiting
  Other Names: anti-emetics

SUMMARY:
* To study the efficacy and side effects of ondansetron with dexamethasone in patients undergoing standard laparoscopic cholecystectomy (control group).
* To study the efficacy and side effects of ramosetron in patients undergoing standard laparoscopic cholecystectomy (study group).
* To compare the efficacy and side effects of ondansetron with dexamethasone and ramosetron in patients undergoing standard laparoscopic cholecystectomy

DETAILED DESCRIPTION:
100 ASA Grade I/II young female patients of 20-40 years undergoing elective laparoscopic cholecystectomy will be equally divided into 2 groups (50 each): control group(Group 'O') and study group (Group 'R') using a computer generated sealed envelopes.

Control group patients will receive ondansetron with dexamethasone and the study group patients will receive ramosetron. Based on the previous studies advocating use of the minimum recommended doses, ramosetron in a dose of 0.3 mg and ondansetron in a dose of 4 mg and dexamethasone in a dose of 8mg will be administered for prevention of PONV in the present study. Medications will be prepared by a blinded paramedic not involved in the study in identical 5-ml syringes and will be administered according to the randomization list. Patients will be given tablet alprazolam(0.25 mg) orally on the night before surgery and advised nil per orally from midnight.

Inside operation theatre, patient NPO status and identity will be reassured. Intravenous line will be secured using 18 G IV cannula and intravenous fluid will be started. Standard non-invasive monitoring will be established intraoperatively using NIBP, HR, ECG, RR, SpO2 and will be continuous postoperatively. Patients will be premedicated with injection Glycopyrrolate (0.004mg/kg), injection Ranitidine (1mg/kg), injection metoclopramide (0.15mg/kg), injection butorphanol (0.04mg/kg). Patients will be induced with injection propofol 2 mg/ kg mixed with xylocard 2%(10mg of xylocard per 10ml propofol) and injection Succinylcholine 1.5 mg/kg and endotracheal intubation will be done. A nasogastric tube will be inserted after securing the endotracheal tube in place and confirming it with ETCO2 monitoring. Anesthesia will be maintained with nitrous oxide and halothane (0.4-1%) in oxygen. Intra-operative muscle relaxation was maintained with injection vecuronium.

At the end of the surgery, injection diclofenac 75 mg IM will be given before the reversal of neuromuscular blockade to pre-empt the post-operative pain and will be advised as IM injection twice a day for post operative analgesia. Additional post-operative analgesia will be provided with injection tramadol 2 mg/ kg slowly as and when required intravenously. Nasogastric suction will be done to remove any residual gastric contents. Residual effect of muscle relaxant will be reversed with injection neostigmine (0.04 mg/ kg) and injection glycopyrrolate (0.2mg for each 1.0 mg 0f neostigmine). Ondansetron (4 mg) with dexamethasone (8mg) or ramosetron (0.3 mg) will be administered intravenously before shifting of the patient from the operation theater to the post-anesthesia care unit (PACU) according to the group allocation. All port sites will be infiltrated with inj bupivacaine (0.25%).

In the post-operative period, patients will be monitored for nausea, vomiting, pain, vital signs, adverse effects and post-anesthetic discharge score for 48 h (every 4 hourly in first 24 hours and every 6 hourly in next 24 hours) and this will be recorded by an independent observer (usually a Resident Officer) who will be blinded to the study. Injection metoclopramide (10 mg I.V.) will be administered as an additional rescue antiemetic in patients with two or more than two episodes of vomiting and/or significant nausea at any time within 48 h of operation. Exact timing of the administration of the rescue antiemetic will be recorded.

Adverse effects of Ramosetron will also be monitored like- Abdominal pain, Hard stools, Constipation, bloating, Hepatic dysfunction, reflux esophagitis, decrease in platelet count, Duodenal ulcer, Palpitation.

Nausea is defined as a subjectively unpleasant sensation associated with awareness of the urge to vomit whereas retching is defined as the labored spasmodic, rhythmic contraction of the abdominal muscles without expulsion of gastric contents, and vomiting is defined as the forceful expulsion of gastric contents from the mouth. Nausea will be measured using an 10 point numerical visual analogue scale with 0 = no nausea and 10 = nausea as bad as can be. A score of > 5 will be considered severe, 5 = moderate and < 5 = minimal. The moderate and severe nausea will be considered as major nausea. During the period of monitoring, the -vomiting/retching episodes of >2 will be considered severe, 2 as moderate, and <2 as mild. Vomiting occurring up to 24 h after surgery will be taken as early vomiting whereas delayed vomiting consist of vomiting occurring during 24-48 h after surgery. A complete response will be defined as the absence of PONV.

ELIGIBILITY:
Inclusion Criteria:

* Female patients of age group 20 - 40years undergoing elective laparoscopic cholecystectomy
* ASA Physical Status- I & II

Exclusion Criteria:

* • Negative consent

  * History of motion sickness
  * Pregnancy
  * Menstruating females
  * Antiemetic taken within 24 hours before surgery or any long term medication
  * History of any systemic diseases, cardio- respiratory, hepato-renal, neurological, endocrinal disorders, hematological disorders, drug or alcohol addiction, psychiatric diseases, study drug sensitivity, etc

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of antiemetic effect of Ramosetron with combination of Ondansetron and Dexamethasone in patients undergoing laparoscopic cholecystectomy | 0-48 hrs post-operative period
  patients will be monitored for vitals, nausea, vomiting, any adverse effect of drug and pain in post-operative period upto 48hrs

CONTACTS AND LOCATIONS:
Locations (1):
- GMC Haldwani, Haldwani, Uttarakhand, India, India

IPD SHARING:
Plan to Share IPD: No